CLINICAL TRIAL: NCT05466266
Title: Comparison of Peri-procedural Complications of Intracardiac Echocardiography and Transesophageal Echocardiography in Patients With Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Sir Run Run Shaw Hospital (Other); Beijing Chao Yang Hospital (Other); First Affiliated Hospital of Suzhou Medical College (Other); Qilu Hospital of Shandong University (Other); RenJi Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Xu Liu, Professor, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ICE VS TEE 2021
Record Dates: First submitted 2021-12-15; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICE group (Experimental): ICE group without TEE detection before procedure
  Interventions: Device: ICE
- TEE group (Active Comparator): TEE group with non-ICE usage at the entire procedure
  Interventions: Device: TEE

INTERVENTIONS:
Device: ICE — All patients received ICE examination.
  Arms: ICE group
Device: TEE — All patients received TEE examination.
  Arms: TEE group

SUMMARY:
Atrial fibrillation (AF) is the most common arrhythmia. Worldwide, the incidence of atrial fibrillation in men and women is 596.2 per 100,000 and 373.1 per 100,000, respectively. [1] The prevalence of AF in China is 0.97%.[2] AF increases the risk of stroke, heart failure and death. Ischemic stroke occurs in 25% of hospitalized patients with nonvalvular atrial fibrillation according to a single-center clinical study in China. [3,4] Complications associated with AF place a huge burden on the healthcare system, with an estimated 4.9 billion RMB for patients with AF in China, 89% of which are caused by AF-related strokes.[5]

According to the 2018 AHA/ACC/HRS guideline [6], catheter ablation was recommended for paroxysmal AF that is symptomatic and refractory or intolerable to at least one class I or III antiarrhythmic drug. Transesophageal echocardiography (TEE) is a necessary preoperative examination for catheter ablation of patients with AF in order to exclude thrombus in the left atrium and left atrial appendage (LAA) and to prevent thrombotic complications caused by thrombus shedding during the procedure. However, TEE detection, like gastroscopy, requires transpharyngeal insertion of the probe into the esophagus and should be fasted before it. The TEE probe is thicker than the gastroscope, which can increase the discomfort of the patient during the examination. At the same time, if the patient cooperates poorly during the delivery process, the probe may damage the oropharyngeal or esophageal mucosa, causing complications such as bleeding or perforation.

Intracardiac echocardiography (ICE) is a new technique that can completely replace TEE in excluding thrombus in left atrium and left atrial appendage. The advantages are that the catheter is inserted from the femoral vein without the discomfort of stimulating the swallowing reflex caused by TEE examination; To avoid complications such as bleeding or perforation caused by injury to oropharynx or esophageal mucosa; It can be used in frail, elderly, pharyngeal or esophageal lesions (eg, ulcers, varices), or intolerable patients. Some studies have shown that ICE is an important test for the diagnosis of LAA thrombosis, especially when thrombus is described as a soft thrombus.

TEE is the gold standard for the detection of thrombi in the LAA before catheter ablation for AF. ICE is used to assist AF ablation; however, ICE is also accurate for LAA visualization and minimizes the complications during procedures[7].

The primary purpose of this study aimed at determining whether ICE could replace TEE by minimizing the procedural-related complications but not compromise the detection of thrombi in the LAA.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-80 years.
2. Willing to sign informed consent.
3. Patients diagnosed with atrial fibrillation Paroxysmal AF and Persistent AF according to the latest clinical guidelines.

Exclusion Criteria:

1. End-stage disease with a mean life expectancy less than 1 year
2. New York Heart Association (NYHA) class III or IV, or last known left ventricular ejection fraction less than 30%
3. Previous surgical or catheter ablation for AF
4. Bradycardia and presence of implanted ICD
5. Uncontrolled hypertension: Systolic blood pressure (SBP) >180 mmHg or diastolic blood pressure (DBP) > 110 mmHg
6. Patients with Cardiovascular events including acute myocardial infarction, any PCI, valvular cardiac surgical, or percutaneous procedure within the past 3 months
7. Women of childbearing potential who are, or plan to become, pregnant during the time of the study
8. Have been enrolled in an investigational study evaluating devices or drugs.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Procedure safety | 18 months
  Procedural-related complications of ICE and TEE.

SECONDARY OUTCOMES:
Thrombus detection rate | 18 months
  Left atrial appendage thrombus detected by ICE and TEE.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu X, Jiang W, Wang X, Ye P, Li X, Wang Y, Zheng Q, Wang Y, Leng L, Zhang Z, Han B, Zhang Y, Qin M, Liu X, Hou X; ICE vs TEE Study Investigators. Intracardiac vs Transesophageal Echocardiography in Atrial Fibrillation Ablation: A Randomized Clinical Trial. JAMA Cardiol. 2025 Dec 1;10(12):1249-1256. doi: 10.1001/jamacardio.2025.3687. PMID 41060665